CLINICAL TRIAL: NCT03224195
Title: Patient Experience of Acute Rehabilitation After Hip Fracture
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 213682
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Hip Fractures; Fracture of Hip; Fractured Hip
Keywords: rehabilitation; patient perspective; semi-structured interview
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore the patient experience of acute rehabilitation after hip fracture surgery. We also aim to identify patient perceived barriers to rehabilitation and recovery after hip fracture surgery. More specifically, the objectives of this study are to:

1. describe the rehabilitation experience of patients who underwent hip fracture surgery with respect to the frequency, intensity, type, and timing of rehabilitation and
2. identify patient perceived barriers to rehabilitation and recovery related to the patient, their injury and their health care.

The results of this qualitative study will inform a future feasibility cluster randomised controlled trial aimed at optimising acute rehabilitation after hip fracture surgery. The findings will help to strengthen the patient and carergiver centred approach when developing the intervention to optimise rehabilitation and potentially improve outcomes after hip fracture surgery.

DETAILED DESCRIPTION:
Each year, UK hospitals admit 75,000 older men and women with fracture of the hip. The injury has been dubbed the "hip attack", due to its clinical severity and adverse consequences. In fact, hip fracture is one of the most detrimental events in an older adult's life. Even with treatment, 30% of patients die within a year.Among survivors, 25% never walk again, and 22% transition from independent living to long-term care. Further, up to one third of patients develop new-onset depressive symptoms post fracture. Many fear admission to a nursing home, in fact a recent study noted that 80% would rather be dead.

Most hip fractures are treated surgically with the goals of reducing pain and re-establishing mobility. Allied health professionals develop rehabilitation interventions targeting the frequency, intensity, type and timing of rehabilitation to improve survival, recovery and quality of life after hip fracture surgery. Evaluation of these interventions rarely offer insight into the patient and caregiver experience. This insight is essential to determine feasibility, acceptability, and ultimately adherence to a new rehabilitation intervention.

As an example, clinicians and researchers suggest the timing of mobilisation will reduce complications and improve recovery after hip fracture surgery, particularly among older patients. The evidence to support these claims is inconsistent. Further, there is limited understanding of the patient experience of early mobilisation after hip fracture surgery. Indeed, for some patients the experience may be improved with a delay to first mobilisation.

To maximise adherence, it is important to also gauge patient's perceptions of perceived barriers to rehabilitation and recovery after hip fracture surgery. These barriers may present in the form of patient characteristics such as motivation. Alternatively, they may present in the form of injury characteristics such as perceived injury severity. Lastly, patient's may perceive healthcare barriers to rehabilitation such as perceived benefit.

DESIGN AND METHODS Design Qualitative study. Semi-structured interview The research assistant will first collect participant demographics - age, sex, previous functional status, previous place of residence - home or long-term care.

Participants will then complete a semi-structured face-to-face interview delivered by a research assistant. The interview will be on an interview topic guide comprised of 3 core topics related to our aims. The questions are flexible, open-ended and broad, while focused on the topic to elicit rich responses from participants. The interviews will explore the experiences of patients who underwent rehabilitation after hip fracture surgery. Each semi-structured interview will last 30-45 minutes and will be recorded with an audio recorder. The research assistant will take reflective field notes to assist interpretation of the interview data.

Data preparation Participant demographics (age, sex, previous functional status, previous place of residence - home or long-term-care) and field notes will be entered into a Microsoft Excel Spreadsheet on a secure controlled access server at Kings College London on the same day as the interview by the research assistant. This server is accessible only to staff at Kings College London. The data will be password-protected and accessible only to the research team.

Recording of semi-structured interviews will be downloaded onto the secure server on the same day as the interview by the research assistant. Recordings will then be permanently deleted from the voice recorder. Interviews will be transcribed verbatim into Microsoft Word documents on the server by the research assistant. Transcripts will then be checked by a Kings College London supervisor, de-identified (by removal of names/locations) and uploaded into the NVivo software. On completion of the transcription the audio recordings will be deleted permanently from the server.

The spreadsheet and transcriptions will be archived on the secure controlled access server for 3 years to allow for analysis, journal submission, response to reviewer's comments, and publication.

Analysis The resulting data will be open coded and thematically analysed using a constant comparative approach with the software package NVivo. Analysis will take place iteratively throughout the project with ongoing coding completed to identify themes and subthemes as they emerge. This will entail the identification of common themes in the data through the reading and re-reading of transcripts first for a descriptive and then an analytic account. Matrices will be used to compare the occurrence of themes across participants.

Upon writing materials for publication, anonymized quotations from the data set will be used to support and illustrate the emergent themes.

Setting George Perkins Ward (trauma orthopaedics), St Thomas's Hospital. The interview will take place in a confidential, private room on the Ward.

Sample size We will recruit 20 participants. We based the sample size on qualitative analysis sample size recommendations. Further, a recent Canadian qualitative study on patient perspective to guide recovery reached data saturation with no new themes emerging after 19 interviews.

Sample technique We will use purposeful-criterion sampling to recruit participants. The first 20 patients/caregivers admitted to George Perkins Ward, St Thomas's Hospital who meet inclusion and exclusion criteria and give informed consent to participate will be included. We chose criterion sampling as we have a predetermined criterion of importance (i.e. adults (and their caregivers) who sustained hip fractures).

Identification of potential participants A member of the clinical team will identify potential participants at the daily multidisciplinary team handover on George Perkins ward, Guy's and St. Thomas' NHS Foundation Trust. During handover, each patient case is discussed including admitting diagnosis, surgery, Abbreviated Mental Test Score (AMTS), functional status, caregiver involvement, and any communication difficulties.

A member of the research team not involved in direct clinical care will be notified by the clinical team of potential participants on attendance at George Perkins Ward. The member of the research team not involved in direct clinical care will then complete the recruitment and consent process.

Recruitment and Consent We will adopt a previous published recruitment strategy developed by the Warwick Hip Trauma Evaluation. As part of usual care patients are assessed for capacity to consent using the 10-item AMTS preoperatively. A score below 8 suggests cognitive impairment.

Those with a score of 8 or more will be approached in hospital after their hip fracture surgery. They (and their caregiver) will be provided with an information sheet and given the opportunity to ask questions. At least 24 hours later they will be given the opportunity to ask any additional questions, and if they wish to take part, to provide written consent. Caregivers who participate will also sign a consent form.

On approach, potential participants and their caregiver will be invited to take part in the study. They will be provided with an information sheet and given the opportunity to ask questions. At least 24 hours later they will be given the opportunity to ask any additional questions, and if they wish to take part, will sign an agreement form and we will aim to interview a caregiver as well as the patient (patient/carer dyad). Caregivers who participate will also sign a consent form.

If the participant declines to participate, we will record the reason offered.

ELIGIBILITY:
Inclusion Criteria:

* • Adult who underwent surgery after admission to St. Thomas's Hospital with hip fracture.

  * Admission during the 9 weeks beginning July 2, 2017.
  * Mobile (with/without aid) before fracture.
  * Informed consent.
  * English speaking.
  * Aged ≥ 60.
  * Abbreviated Mental Test Score ≥ 8/10.

Exclusion Criteria:

* • Adults who do not undergo surgery after admission to St. Thomas's Hospital with hip fracture.

  * Admissions outside the 9 weeks beginning July 2, 2017.
  * Not mobile before fracture.
  * Aged< 60.
  * Not English speaking.
  * AMTS < 8/10.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged 65 and over who have been admitted for surgical management of hip fracture who were mobile prior to fracture and do not have cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
patient perspective of acute rehabilitation following hip fracture | interviews over 8 weeks
  nil outcome measure- semi-structured interview

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom